CLINICAL TRIAL: NCT05597423
Title: Massage as a Recovery Strategy After Resistance Training: Randomized Clinical Trial
Brief Title: Massage as Recovery Strategy After Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Flávia Carvalho, Principal investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECM_22
Record Dates: First submitted 2022-10-15; First posted 2022-10-28 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Resistance Training
Keywords: Massage; Physical activity; Perception; Recovery
MeSH Terms: conditions — Motor Activity | interventions — Massage

STUDY DESIGN:
Intervention Model Description: All interventions will take place 10 minutes after the end of resistance training focused on the lower limbs (twice a week for four weeks). The intervention group will receive the massage for 16 minutes in 4 muscle groups bilaterally: i) quadriceps ii) calf iii) hamstrings iv) lower back. The techniques used will be the superficial effleurage followed by the deep effleurage, petrissage and tapotement. In the placebo group, the same cream used to perform the massage will be spread over the quadriceps, calf, hamstrings and lower back with three superficial slides on each musculature to spread the cream. This process will be carried out bilaterally and the participant will be asked to remain in the supine position for 16 minutes. In the control group, participants will be asked to rest for 16 minutes and the participants can be seated, standing or walking through the space during this period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage (Experimental): The massage will be applied twice a week for a period of four weeks, 10 minutes after the end of lower limb training.
  Interventions: Other: Massage
- Placebo (Placebo Comparator): The massage cream will be applied twice a week for a period of four weeks, 10 minutes after the end of lower limb training.
  Interventions: Other: Placebo
- Control (No Intervention): The control group after 10 minutes of the end of lower limb training will remain at rest for 16 minutes.

INTERVENTIONS:
Other: Massage — The massage will be applied for 16 minutes on the quadriceps, calf, hamstrings and lower back bilaterally with 4 different pressures.
  Arms: Massage
Other: Placebo — The cream will be applied to the quadriceps, calf, hamstring and lower back bilaterally and the participant will wait 16 minutes lying down in the supine position.
  Arms: Placebo

SUMMARY:
Within the routine of resistance training, stimulus are implemented to meet predetermined goals for its practitioners. In order for there to be a balance in the imposed loads, a recovery period is necessary for supercompensation to occur. Recovery is a multifactorial process and to consider an individual recovered it is necessary to respect the integration of physiological, biomechanical and psychological factors, in addition, perceptual markers, which are not widely investigated in the literature, seem to be effective recovery markers. Massage is a technique that stands out for its wide use after physical exercise in order to help accelerate the recovery process. In the literature, studies that investigated the influence of massage on performance did not find positive results and some authors question the real need to apply the technique to aid recovery. However, in the perceptual parameters, massage seems to have a good influence, such as pain reduction, perception of fatigue and improvement in the perception of recovery. Thus, understanding the experience that massage can provide during a training period can be an important outcome along with variables already used. The hypothesis of this study is that massage will improve perceptual parameters over a training period and, consequently, will improve the experience between training sessions without positively or negatively interfering in performance.

DETAILED DESCRIPTION:
A sample of 120 participants will be recruited for the study. This is a parallel randomized controlled clinical trial lasting 4 weeks, each week will consist of 5 resistance training sessions. Participants will be randomized into three groups, control, intervention or placebo. Interventions will take place after training focused on the lower limbs. The intervention group will receive a massage for 16 minutes, in the placebo group the massage cream will be applied and the participants will be asked to remain in the supine position for 16 minutes and the control group will wait the same time at rest. All participants will perform an initial assessment consisting of an initial screening questionnaire, referred morbidity index, jump test and strength test. At the beginning, during and at the end of each lower limb training, after the interventions over 96 hours, the perceptual parameters will be evaluated and the assessment of muscle tone and stiffness, elasticity, mechanical stress relaxation time and creep will be before and after the training and after the intervention. On the second day of the lower limb training on each week, the Squat Jump Test will be evaluated before, after training and after the intervention. At the end of the 4 weeks of training, the participant will perform evaluations of functional and strength outcomes. At the end of the study, the preference of the participant and the cost-benefit of the technique will also be evaluated. Participant satisfaction will be evaluated after the technique. At the end of each week and at the end of the study, a balance of outcomes will be carried out. At the end of the study, the participant will also answer a questionnaire about sensations during training to perform a qualitative analysis. Data will be described as mean and standard deviation or median and interquartile range depending on the data distribution. Data normality will be tested by the Shapiro-Wilk test. Comparisons between techniques and associations will be performed using generalized mixed models with post Bonferroni test. All analyzes will assume a significance level of p>0.05.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 35 years;
* practice resistance training for at least 2 months;
* train at least 5 times a week;
* not having suffered an injury in the last 6 months in the lower limbs;
* not being a smoker.

Exclusion Criteria:

* use anti-inflammatory and/or analgesic medication during the study period;
* present an inflammatory process during the study period;
* not reaching 80% frequency in lower limb training during the study period.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Perceptual parameters | Up to 4 weeks before all lower limb training
  Post-Exercise Perception Questionnaire (topic before training). The questionnaire will assess the following perceptual parameters: well-being, physically prepared for training, mentally prepared for training, perception of mental fatigue, lower limb fatigue, lower limb muscle pain, sensation of lower limb muscle tension, lower limb muscle discomfort and perception of recovery. All parameters will be evaluated by a 5-point Likert scale (1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely)
Perceptual parameters | Up to 4 weeks during all lower limb training
  Post-Exercise Perception Questionnaire (topic during training). The questionnaire will assess the following perceptual parameters: lower limb fatigue, lower limb muscle pain, sensation of lower limb muscle tension and lower limb muscle discomfort. All parameters will be evaluated by a 5-point Likert scale (1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely)
Perceptual parameters | Up to 4 weeks after all lower limb training
  Post-Exercise Perception Questionnaire (topic after training). The questionnaire will assess the following perceptual parameters: well-being, perception of mental fatigue, lower limb fatigue, lower limb muscle pain, sensation of lower limb muscle tension, lower limb muscle discomfort and perception of recovery. All parameters will be evaluated by a 5-point Likert scale (1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely)
Perceptual parameters | Up to 4 weeks after the application of intervention in all lower limb training
  Post-Exercise Perception Questionnaire (topic after training). The questionnaire will assess the following perceptual parameters: well-being, perception of mental fatigue, lower limb fatigue, lower limb muscle pain, sensation of lower limb muscle tension, lower limb muscle discomfort and perception of recovery. All parameters will be evaluated by a 5-point Likert scale (1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely)
Perceptual parameters | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1, 2, 4, 8, 12, 16, 20, 24, 48, 72 and 96 hours after the application of intervention in all lower limb training up to 4 weeks
  Post-Exercise Perception Questionnaire (topic between trainings). The questionnaire will assess the following perceptual parameters: well-being, lower limb fatigue, lower limb muscle pain, sensation of lower limb muscle tension, lower limb muscle discomfort and perception of recovery. All parameters will be evaluated by a 5-point Likert scale (1=nothing; 2= a little; 3=moderate; 4=a lot; 5=extremely)

SECONDARY OUTCOMES:
Inferior limb power | Change from baseline to 4 weeks
  Inferior limb power will be measured by the squat jump test (cm)
Inferior limb power | Up to 4 weeks change from baseline to after lower limb training
  Inferior limb power will be measured by the squat jump test (cm)
Inferior limb power | Up to 4 weeks change from baseline to after the application of intervention in lower limb training
  Inferior limb power will be measured by the squat jump test (cm)
Lower limb strength | Change from baseline to 4 weeks
  Lower limb strength will be measured by the one-repetition maximum test
Muscle tone | Up to 4 weeks change from baseline to after all lower limb training
  Muscle tone will be measured in hertz by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Muscle tone | Up to 4 weeks change from baseline to after the application of intervention in all lower limb training
  Muscle tone will be measured in hertz by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Muscle stiffness | Up to 4 weeks change from baseline to after all lower limb training
  Muscle stiffness will be measured in newton meter by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Muscle stiffness | Up to 4 weeks change from baseline to after the application of intervention in all lower limb training
  Muscle stiffness will be measured in newton meter by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Elasticity | Up to 4 weeks change from baseline to after all lower limb training
  Elasticity will be measured in logarithmic decrement of natural oscillation (logD) by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally
Elasticity | Up to 4 weeks change from baseline to after the application of intervention in all lower limb training
  Elasticity will be measured in logarithmic decrement of natural oscillation (logD) by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally
Mechanical stress relaxation time | Up to 4 weeks change from baseline to after all lower limb training
  Mechanical stress relaxation time will be measured in milliseconds by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Mechanical stress relaxation time | Up to 4 weeks change from baseline to after the application of intervention in all lower limb training
  Mechanical stress relaxation time will be measured in milliseconds by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Creep | Up to 4 weeks change from baseline to after all lower limb training
  Creep (relationship between relaxation time and muscle deformation time) will be measured by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally.
Creep | Up to 4 weeks change from baseline to after the application of intervention in all lower limb training
  Creep (relationship between relaxation time and muscle deformation time) will be measured by the MyotonPRO device wich has a probe that will be placed perpendicular to the skin surface on the muscle belly previously marked with a pen by the evaluator at the quadriceps, hamstrings, lumbar multifidus and soleus bilaterally
Technical preference | Week 4
  The participant will be asked about the preference of the technique included in the training routine (yes or no)
Technique belief | Week 4
  Participants will answer how they believe the technique is cost-effective using a 5 point likert scale (1=poor, 2=bad, 3=indifferent, 4=good, 5=excellent)
Participant satisfaction about the technique assessed by a 5-point Likert scale [followed by its scale information in the Description] | Up to 4 weeks immediately after intervention
  The participant will be asked about satisfaction of the technique received using a 5 point likert scale (1=completely dissatisfied, 2=dissatisfied, 3=neither satisfied nor dissatisfied, 4=satisfied, 5=completely satisfied)
Participant's perception of the training | Week 4
  Participants will be asked to answer the open questions for a qualitative analysis: "What positive and/or negative feelings do you have after an lower limb training? Describe how they appear or develop over time, including your activities of daily living.", " Considering the recovery strategy used for you after your lower limb training, talk about: how do you feel during this moment? What do you believe that what is done during this period gives you in relation to recovery? Your preference regarding what to do immediately after training." and "Are there any sensations related to the training you perform that you would like to eliminate? What would they be and would you invest time and/or money to eliminate them?"

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Pastre, PhD, Study Director — São Paulo State University
Locations (1):
- Sao Paulo State University, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No